CLINICAL TRIAL: NCT01415830
Title: Randomized Controlled Trial To Evaluate Efficacy And Safety Of The Polyvalent Anti-scorpion Venom Serum Of Birmex Versus Other Commercial Venom Serum In Children Population
Brief Title: Compare Two Anti-Scorpion Venom Serum In Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratorios de Biologicos y Reactivos de México, S.A. de C.V. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: BIRMEX-ECA-03-2011
Record Dates: First submitted 2011-08-08; First posted 2011-08-12 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Scorpion Sting
Keywords: Anti-Scorpion venom serum; venom; efficacy; safety; children
MeSH Terms: conditions — Scorpion Stings

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anti-scorpion venom serum Birmex (Experimental): Patients 0 to 15 years with scorpion sting, will receive serum antiscorpion elaborated by Birmex
  Interventions: Biological: Anti-scorpion venom serum Alacramyn
- Anti-scorpion venom serum Alacramyn (Active Comparator): Patients 0 to 15 years with scorpion sting, will receive other commercial serum antiscorpion (Alacramyn)
  Interventions: Biological: Anti-scorpion venom serum Birmex

INTERVENTIONS:
Biological: Anti-scorpion venom serum Birmex — the dose may be required for the patient according to clinical manifestations and evolution
  Other Names: anti-scorpion venom serum
  Arms: Anti-scorpion venom serum Alacramyn
Biological: Anti-scorpion venom serum Alacramyn — The dose may be required fot the patient according to clinical manifestations and evolution
  Other Names: antiscorpion venom serum
  Arms: Anti-scorpion venom serum Birmex

SUMMARY:
The morbidity associated with scorpion sting intoxication presents an endemic pattern in the country, where there are highly venomous species of scorpions so the scorpion sting intoxication (IPPA) is considered a medical emergency.

On the other hand, there is scarce scientific literature from different controlled studies evaluating anti-scorpion serum, considering clinical severity scales, lab results and their safety. The aim of this study is to compare the efficacy and safety of scorpion sting treatment, using two sera, one produced by Birmex versus Alacramyn ® (Bioclon).

DETAILED DESCRIPTION:
We consider relevant conduct this study because the poisoning scorpion bite represents a public health problem.

This is a randomized clinical trial, which included 120 subjects of both sexes aged 0 and 15 years old and residents of the state of Guanajuato, divided into 2 groups: 60 patients received antiscorpion serum of Birmex and 60 patients receive other commercial serum (Alacramyn).

ELIGIBILITY:
Inclusion Criteria:

1. Scorpion sting
2. Either sex
3. Age 1 to 15 years
4. Signing an informed consent (signed by parent or guardian)
5. Being residents of the state of Guanajuato

Exclusion Criteria:

1. Previous treatment with gamma globulin or immunoglobulin
2. Blood transfusion at any stage of life
3. Patients treated with drugs that interact with anti-scorpion serum
4. History or history of sensitivity or intolerance to anti-scorpion serum or horse products
5. Pregnancy
6. Any immunodeficiency
7. Patients who have participated in a research protocol in the previous month.

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2011-08; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Resolution of signs and symptoms of scorpion envenomation | after treatment (expected average of 12 hrs)

SECONDARY OUTCOMES:
Evaluate the adverse events in every treated child | inmediately after treatment and until 5 days later

CONTACTS AND LOCATIONS:
Overall Officials: Ma. Eugenia Jimenez-Corona, PhD, Principal Investigator — Laboratorios de Biologicos y Reactivos de México SA de CV
Locations (1):
- Hospital General Regional de León, León, Guanajuato, Mexico